CLINICAL TRIAL: NCT00705224
Title: Observational Multicenter Study to Evaluate Influence of Insulin Resistance on the Safety and Efficacy (as Measured by Sustained Virological Response) of Treatment With Any Pegylated Interferon and Ribavirin (Standard of Care) in Different Populations of HCV Patients in Russia.
Brief Title: Effect of Insulin Resistance on the Safety and Efficacy of Pegylated Interferon and Ribavirin Treatment in HCV (Study P05562)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05562
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C, Chronic; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis C: Naïve patients with chronic hepatitis C (CHC) of any genotype will be treated with a standard treatment regimen (pegylated interferon and ribavirin) according to routine clinical practice in Russia.
  Interventions: Biological: Pegylated Interferon; Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated Interferon — Routine treatment with a combination of any pegylated interferon and ribavirin was used according to the label/local practice in Russia.
  The treatment course duration complied with the labeled dosage regimen. Each dose of pegylated interferon was administered as a subcutaneous
  injection calculated as 1.5 mcg/kg once a week. Therapy duration varied from 24 to 48 weeks depending on Hepatitis C virus (HCV) genotype, viral load, activity and stage of hepatitis C.
  The Sponsor did not provide formal drug supply.
  Other Names: PegIntron; (SCH 54031)
Drug: Ribavirin — Routine treatment with a combination of any pegylated interferon and ribavirin was used according to the label/local practice in Russia.
  The treatment course duration complied with the labeled dosage regimen. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the
  morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and stage of hepatitis C.
  The Sponsor did not provide formal drug supply.
  Other Names: Rebetol; (SCH 18908)

SUMMARY:
Naïve patients with chronic hepatitis C (CHC) of any genotype will be treated with a standard treatment regimen (pegylated interferon and ribavirin) according to routine clinical practice in Russia. The objective of this study is to examine the influence of insulin resistance on the safety and efficacy of treatment with pegylated interferon and ribavirin and to determine the prevalence of insulin resistance in different populations of CHC patients.

DETAILED DESCRIPTION:
consecutive patient sampling

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CHC according to local regulations
* Naïve Pegylated Interferon (PEG-IFN) CHC patient
* No contraindications for PEG-IFN CHC therapy
* Negative urine pregnancy test result (for females of childbearing potential) documented within the 24-hour period prior to the first dose of study drugs. Additionally, all female patients of childbearing potential and all males with female partners of childbearing potential must use two forms of effective contraception (combined) during treatment and 6 months after treatment end
* Willingness to give written informed consent and willingness to participate in and comply with the study requirements.

Exclusion Criteria:

* PEG-IFN treatment in history
* Contraindications for PEG-IFN CHC therapy
* Females who are pregnant or breast-feeding
* Male partners of females who are pregnant
* Potentially unreliable participants, and those judged by the investigator to be unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include naïve patients with chronic hepatitis C (CHC) of any genotype who will be treated with a standard treatment regimen (pegylated interferon and ribavirin) according to routine clinical practice in Russia.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated Interferon and Ribavirin: Naïve patients with chronic hepatitis C (CHC) of any genotype treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous
  injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the
  morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on hepatitis C virus (HCV) genotype, viral load, activity and stage of hepatitis C.
Period: Overall Study
Arm/Group | Pegylated Interferon and Ribavirin
Started | 250
Completed | 239
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Pegylated Interferon and Ribavirin: Naïve patients with CHC of any genotype treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous
  injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the
  morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and stage of hepatitis C.
Arm/Group | Pegylated Interferon and Ribavirin
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 146

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sustained Virological Response as Assessed at End of Study
Description: Sustained Virological response (SVR) was assessed at the end of the study (Visit 4) to investigate the presence or absence of SVR. SVR was defined as undetectable plasma hepatitis C virus RNA (HCV-RNA) at 24 weeks after termination of treatment. Visit 4 was considered Week 48 or Week 72 depending on a treatment duration of 24 or 48 weeks respectively.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Completer set for the primary analysis included all participants who were administered at least one dose of the study treatment and provided the SVR data at end of study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pegylated Interferon and Ribavirin
Number analyzed (Participants) | 223
Percentage of Participants | 81.2 [76.0 to 86.3]

2. Secondary Outcome: Percentage of Participants Who Achieved Sustained Virological Response as Assessed at End of Study by HCV Genotype and Presence of Insulin-Resistance at Baseline
Description: SVR was assessed at the end of the study (Visit 4) by HCV genotype (I, II, III, or other) and presence of insulin-resistance at baseline (defined as Homeostasis model assessment - of insulin-resistance [HOMA-IR] >3) to investigate the presence or absence of SVR. SVR was defined as undetectable plasma HCV-RNA at 24 weeks after termination of treatment. Visit 4 was considered Week 48 or Week 72 depending on a treatment duration of 24 or 48 weeks respectively.
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Completer set for the primary analysis (N=223) included all participants who were administered at least one dose of the study treatment and provided the SVR data at end of study. Of the 223 participants in this population, 181 achieved SVR (N=140 and N=40) and were therefore included in this analysis. 1 participant of the 181 had missing values.
Measure: Number; unit: Percentage of Participants
Groups:
- HOMA-IR<=3: Subgroup of naïve patients with CHC of any genotype and an absence of insulin resistance at baseline treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and stage of hepatitis C.
- HOMA-IR >3: Subgroup of naïve patients with CHC of any genotype and a presence of insulin resistance at baseline treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and stage of hepatitis C.
Arm/Group | HOMA-IR<=3 | HOMA-IR >3
Number analyzed (Participants) | 140 | 40
Percentage of Participants
  Genotype I | 45.7 | 47.5
  Genotype II | 14.3 | 7.5
  Genotype III | 38.6 | 45.0
  Other | 1.4 | 0

3. Secondary Outcome: Percentage of Participants Who Achieved Response Following Treatment as Assessed at End of Treatment by HCV Genotype and Presence of Insulin-Resistance at Baseline
Description: Response following treatment (RFT) was assessed at the end of treatment (Visit 3) by HCV genotype (I, II, III, or other) and presence of insulin-resistance at baseline (defined as HOMA-IR >3) to investigate the presence or absence of RFT. RFT was defined as undetectable plasma HCV-RNA at end of treatment. Visit 3 was considered Week 24 or Week 48 after treatment start depending on treatment duration.
Time Frame: Week 24 or 48 after treatment start
Population: Completer set for the primary analysis (N=223) included all participants who were administered at least one dose of the study treatment and provided the SVR data at end of study. Of the 223 participants in this population, 208 achieved RFT (N=156 and N=51) and were therefore included in this analysis. 1 participant of the 208 had missing values.
Measure: Number; unit: Percentage of Participants
Arm/Group | HOMA-IR<=3 | HOMA-IR >3
Number analyzed (Participants) | 156 | 51
Percentage of Participants
  Genotype I | 50.6 | 52.9
  Genotype II | 12.2 | 5.9
  Genotype III | 35.9 | 41.2
  Other | 1.3 | 0

4. Secondary Outcome: Percentage of Participants Who Demonstrated Virological Relapse as Assessed at End of Study by HCV Genotype and Presence of Insulin-Resistance at Baseline
Description: Virological relapse (VR) was assessed at the end of the study (Visit 4) by HCV genotype (I, II, III, or other) and presence of insulin-resistance at baseline (defined as HOMA-IR >3) to investigate the percentage of participants who demonstrated VR. VR was defined as undetectable plasma HCV-RNA (RFT +) at end of treatment (Visit 3- considered Week 24 or Week 48 after treatment start depending on treatment duration), but lost RFT (considered sustained non-Responders) at end of study (Visit 4- considered Week 48 or Week 72 depending on a treatment duration of 24 or 48 weeks respectively).
Time Frame: 24 weeks following completion of 24 or 48 weeks of therapy
Population: Completer set for the primary analysis (N=223) included all participants who were administered at least one dose of the study treatment and provided the SVR data at end of study. Of the 223 participants in this population, 29 participants demonstrated virological relapse (N=18 and N=11) and were therefore included in this analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- HOMA-IR<=3: Subgroup of naïve patients with CHC of any genotype and an absence of insulin resistance at baseline treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and a stage of hepatitis C.
Arm/Group | HOMA-IR<=3 | HOMA-IR >3
Number analyzed (Participants) | 18 | 11
Percentage of Participants
  Genotype I | 83.3 | 72.7
  Genotype II | 0 | 0
  Genotype III | 16.7 | 27.3
  Other | 0 | 0

5. Secondary Outcome: Percentage of Participants Who Achieved Early Virological Response as Assessed at Visit 2 by HCV Genotype and Presence of Insulin-Resistance at Baseline
Description: Early Virological response (EVR) was assessed at 12 weeks after treatment start (Visit 2) by HCV genotype (I, II, III, or other) and presence of insulin-resistance at baseline (defined as HOMA-IR >3) to investigate the percentage of participants who achieved EVR. EVR was defined as a substantial (greater than 2 log10) decrease in viral load (measured as International Units/milliliter) and/or negative Polymerase chain reaction (PCR)-based viral load qualitative result as assessed at visit 2 of the study.
Time Frame: Week 12 after treatment start
Population: Completer set for the primary analysis (N=223) included all participants who were administered at least one dose of the study treatment and provided the SVR data at end of study. Of the 223 participants in this population, 210 participants demonstrated early virological response (N=158 and N=50). 2 participants of the 210 had missing values.
Measure: Number; unit: Percentage of Participants
Arm/Group | HOMA-IR<=3 | HOMA-IR >3
Number analyzed (Participants) | 158 | 50
Percentage of Participants
  Genotype I | 51.3 | 54.0
  Genotype II | 12.7 | 6.0
  Genotype III | 34.8 | 40.0
  Other | 1.3 | 0

ADVERSE EVENTS:
Description: Safety set: All participants who were administered at least one dose of the study treatment.
Groups:
- Pegylated Interferon and Ribavirin: Naïve patients with chronic hepatitis C (CHC) of any genotype treated with a standard treatment regimen of pegylated interferon and ribavirin according to routine clinical practice in Russia. Each dose of pegylated interferon was administered as a subcutaneous
  injection calculated as 1.5 mcg/kg once a week. The doses were corrected in case adverse events related to pegylated interferon registered. Ribavirin was taken orally as 200 mg gelatinous capsules. The daily dose varied from 800 to 1200 mg (depending on patient's body weight) twice daily in the
  morning and in the evening with meal. Therapy duration varied from 24 to 48 weeks depending on HCV genotype, viral load, activity and stage of hepatitis C.
Arm/Group | Pegylated Interferon and Ribavirin
Serious Adverse Events (participants affected / at risk) | 2/250
Other Adverse Events (participants affected / at risk) | 177/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon and Ribavirin (N=250)
Drug Exposure During Pregnancy (Injury, poisoning and procedural complications) | 1 (1)
Acoustic Neuritis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon and Ribavirin (N=250)
Anaemia (Blood and lymphatic system disorders) | 69 (69)
Leukopenia (Blood and lymphatic system disorders) | 90 (90)
Neutropenia (Blood and lymphatic system disorders) | 30 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 50 (50)
Asthenia (General disorders) | 31 (31)
Influenza Like Illness (General disorders) | 91 (91)
Pyrexia (General disorders) | 17 (17)
Weight Decreased (Investigations) | 26 (26)
Depression (Psychiatric disorders) | 25 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees for a period of five years following the Effective Date to retain the Disclosure made to the SPONSOR or on behalf of SPONSOR, in confidence and not disclose it to any third party.